CLINICAL TRIAL: NCT06543745
Title: Safety and Impact of Low Resistance Exercise Training on Quality of Life in Pulmonary Arterial Hypertension
Acronym: RESIST-PH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 855504
Record Dates: First submitted 2024-06-20; First posted 2024-08-09 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Pulmonary Arterial Hypertension; Frailty
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subjects (Experimental): All subjects will participate in the low-resistance training
  Interventions: Behavioral: Low-Resistance Training

INTERVENTIONS:
Behavioral: Low-Resistance Training — The following 6 exercises will be performed in 3 sets of 15-15-15 repetitions, 3 times per week for 12 weeks:
  Elbow Flexion, Elbow Extension, Lateral Hip Extensions, Hip Extensions, Knee Extensions, Wall push-ups

SUMMARY:
The purpose of the study is to learn more about how low-resistance training impacts frailty and the quality of life of people with pulmonary arterial hypertension (PAH). Low-resistance training is an evidence-based approach that may help patients improve their functional ability.

DETAILED DESCRIPTION:
Patients with pulmonary arterial hypertension and their caregivers will be asked to participate in the study. The study consists of a baseline in-person visit (week 1) where quality of life and physical performance will be assessed, and subjects will be shown low-resistance training exercises to perform at home. The exercises will then be performed at home, as instructed, for 12 weeks. At week 12, subjects return for a follow-up in-person visit, where quality of life and physical performance will be reassessed. Patients and caregivers will also be asked to participate in separate exit interviews, where investigators will ask how they felt about the resistance training.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PAH: idiopathic, heritable, associated with connective tissue disease, congenital heart disease, human immunodeficiency virus, drug- or toxin, or portopulmonary hypertension
* On stable PAH therapy for 3 months

Exclusion Criteria:

* World Health Organization (WHO) functional class IV
* Left ventricular ejection fraction < 40% (via transthoracic echocardiogram (TTE) within one year of screening)
* Moderate or severe concomitant lung disease: Chronic Obstructive Pulmonary Disease (COPD) or interstitial lung disease
* Enrollment in a clinical trial
* Recent hospitalization (within 4 weeks of screening)
* Inability to perform the Short Physical Performance Battery or wheelchair bound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Between baseline and 12-week follow-up
  Safety will be assessed by way of the incidence of serious adverse events.
Feasibility of Recruitment | Through study completion, an average of twice per year
  Feasibility of recruitment will be assessed by measuring recruitment rates
Feasibility of Study | Through study completion, an average of twice per year
  Feasibility of the study will be assessed by measuring retention rates.
Short Performance Physical Battery (SPPB) and emPHasis-10 (E10) scores | Between baseline and 12-week follow-up
  Investigators will use a change in score for SPPB and E10 scores, using Wilcoxon signed-rank test.
Patient/ Caregiver Exit Interview | Upon conclusion of the 12-week follow-up
  Each subject (both patients who participate in the study and their caregivers, separately) will be asked to review their experience with the study protocol, rating their satisfaction on a 5 point Likert scale (1 being Strongly Disagree, 5 being Strongly Agree) with the overall protocol, ease of exercises, acceptability of equipment and exercises. Higher scores (eg. agreement of a positive experience) mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Al-Naamani, MD, MS, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsyvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-04-09): https://cdn.clinicaltrials.gov/large-docs/45/NCT06543745/ICF_000.pdf